CLINICAL TRIAL: NCT04626206
Title: Multi-paramEtric Imaging to Assess Treatment REsponse After Stereotactic Radiosurgery of Brain Metastases
Brief Title: Multi -paramEtric Imaging to Assess Treatment REsponse After Stereotactic Radiosurgery of Brain Metastases
Acronym: METRE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: CCR5331
Record Dates: First submitted 2020-11-03; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Brain Metastases, Adult
Keywords: brain metastases; stereotactic radiosurgery; multi-parametric MRI; contrast-clearance analysis MRI; TRAMs; 18F-choline PET/CT; treatment response
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Imaging to asess treatment response post-SRS: There will be only one group. All recruited patients will have 3 scans, the multi-parametric MRI, contrast-clearance analysis MRI (TRAMs) and 18F-choline-PET/CT.
  This is a non interventional study. Only the results of the contrast-clearance analysis MRI (TRAMs) will be used to make clinical decisions (as this is the current standard of care at the recruiting site). The multi-parametric MRI and 18F-choline PET/CT will be treated as research scans.

SUMMARY:
After stereotactic radiosurgery (SRS) of brain metastases, patients undergo a standard brain magnetic resonance imaging (MRI) to assess treatment response 12 weeks after completion of treatment. The interpretation of this standard MRI can sometimes be challenging as it can be difficult to differentiate tumour getting bigger/returning (progression/recurrence) from expected radiotherapy treatment-related changes known as radionecrosis. This study is a pilot brain imaging study that is investigating if readily available forms of imaging such as contrast-clearance analysis MRI (also known as TRAMs) and/or 18 Fluoromethyl-choline positron emission tomography/computerised tomography (18F-choline PET/CT) are equivalent to multi-parametric MRI in their ability to differentiate tumour from radionecrosis. Multi-parametric MRI has the most evidence for its ability to discriminate tumour from radionecrosis but is resource intensive and not routinely available in most centres.

DETAILED DESCRIPTION:
Differentiating tumour progression/recurrence from radionecrosis post- stereotactic radiosurgery (SRS) of brain metastases can be at times challenging on standard brain MRI. This is because radionecrosis mimics the appearances of tumour progression by appearing as contrast enhancing lesions on standard MRI.The definitive way of differentiating this is surgical excision of the area in question and histopathological evaluation. But this is not always feasible in clinical practice as not all areas of the brain are surgically accessible and an en bloc (complete) resection is needed for the result to be meaningful.

The next best option we have is the multi-parametric MRI which typically consists of three components-MR perfusion, MR diffusion and MR spectroscopy. This investigation is resource intensive, requiring considerable input form MR physics, neuroradiology reporting time , is not routinely available in all centres and hence not viable for routine clinical practice.

Therefore there is an urgent need for a reliable and viable form of imaging modality that helps differentiate tumour from radionecrosis when assessing treatment response post-SRS. It is important to be able to do this accurately as the management of both conditions are entirely different.

Currently the Royal Marsden Hospital is using contrast-clearance analysis MRI (TRAMs) to help differentiate tumour from radionecrosis if the changes seen on standard brain MRI post-SRS are deemed to be unclear. Contrast-clearance analysis MRI (TRAMs) is FDA approved and conforms to European standards (CE marked), yet has sparse evidence on its efficacy. There is some evidence for the use of 18F-choline PET/CT in primary brain tumours (gliomas) but more evidence is needed for its use in brain metastases.

Given that surgical excision is not always feasible for reasons explained above, in this study the investigators consider the muti-parametric MRI as the gold standard investigation for discriminating tumour from radionecrosis.

This pilot brain imaging study is seeking to determine if contrast-clearance analysis MRI (TRAMs) and/or 18F-choline PET/CT are equivalent to multi-parametric MRI in their ability to reliably differentiate between tumour progression/recurrence and radionecrosis. If contrast clearance analysis MRI (TRAMs) and/or 18F-choline PET/CT are found to be equivalent to multi- parametric MRI then it gives the investigators increased confidence in the findings of these readily available imaging modalities, helping treating clinicians to make rapid and reliable management plans- ultimately improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain metastases whose primary cancer originates from the lung and whose histology is that of non-small cell lung cancer (NSCLC)
* Patient should have had SRS as their primary treatment for their brain metastases
* Follow-up standard brain MRI post-SRS has been discussed in the SRS multi-disciplinary team meeting (MDT)
* The changes seen on the post-SRS follow-up standard MRI are deemed unclear by the SRS MDT as to whether they represent tumour progression or radionecrosis.
* It is >=12 weeks since completion of SRS

Exclusion Criteria:

* Prior SRS or external beam radiotherapy to the same area
* Children (age < 18)
* Pregnant women
* Adults that lack capacity to consent
* Contraindications to intravenous gadolinium contrast and/or 18F-choline radiotracer
* Contraindications to MRI scanning (for example pacemaker )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients with brain metastases who have undergone primary stereotactic radiosurgery for their brain metastases. These patients have had a follow up standard brain MRI to assess treatment response and this has been discussed in the stereotactic radiosurgery multidisciplinary team meeting (MDT) and the MDT has deemed that the changes seen are unclear as to whether they represent tumour progression or radionecrosis.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Equivalence of the contrast-clearance analysis MRI (TRAMs) and/or 18F-Choline PET/CT to multi-parametric MRI in differentiating tumour progression/recurrence from radionecrosis post stereotactic radiosurgery of brain metastases. | Primary outcome will be measured after the last visit of last patient-about 8 months from first recruited patient.
  Patients will be classified into two groups according to the result of each scan with either tumour progression/recurrence or radionecrosis (i.e. tumour or no tumour).
  Patients will have all three scans within two weeks of each other, and then each imaging technique will be reviewed and reported by neuroradiologists as either disease or no disease. All three scans will be assessed once.
  The sensitivity, specificity, positive and negative predictive values in detecting tumour and prevalence will be calculated for the two scan methods where multi-parametric MRI will be used as the definitive diagnosis as we consider this as the gold standard in this study. The two scan methods are contrast-clearance analysis MRI (TRAMs) and 18F-choline PET/CT classification (tumour or no tumour) which will be compared against multi-parametric MRI. These separate measurements will be aggregated to obtain the primary outcome measurement (equivalence).

SECONDARY OUTCOMES:
Secondary endpoints are exploratory and will focus on correlating quantitative imaging derived parameters from contrast-clearance analysis MRI (TRAMs) and 18F-choline PET/CT with quantitative parameters in multi-parametric MRI. | This can be measured after the last visit of last patient-about 8 months from first recruited patient.
  Each imaging technique, multi-parametric MRI (this scan has 3 components), contrast-clearance analysis MRI (TRAMs) and 18F-choline PET, measures different quantitative parameters to assess for the presence of tumour. Examples of quantitative parameters include for multi-parametric MRI: relative cerebral blood volume, apparent diffusion coefficient, choline to n-acetylcysteine ratio; contrast-clearance analysis MRI (TRAMs): volume of red versus blue areas on the treatment assessment maps; 18F-Choline PET: uptake value of the 18F-choline. These separate measurements will be aggregated to measure a single outcome, outcome 2 which is - is there a correlation between quantitative parameters from TRAMs and 18F-choline PET/CT and multi-parametric MRI.
Correlation of the three scan results with the actual clinical outcomes for the patients-ie tumour or radionecrosis. | Analysed only after a follow-up period of at least 6 months for all patients post completion of study investigations-about 14 months from first recruited patient and 6 months from last recruited patient.
  Results from the three imaging modalities contrast-clearance analysis MRI (TRAMs), 18F-choline PET/CT, multi-parametric MRI, will be compared with the actual clinical outcomes for the patients (i.e. tumour progression/recurrence or radionecrosis) which will be known with more certainty after a period of follow-up of 6 months has elapsed following the study imaging investigations. This follow-up involves collecting routine standard brain MRI scan results (reports and/or images) and clinical review letters from the primary team.
  The sensitivity, specificity, positive and negative predictive values in detecting tumour and prevalence for the three scan methods will be compared against actual clinical outcomes. These separate measurements will be aggregated to measure outcome 3, which is - is there a correlation between the three scans and actual clinical outcomes for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Liam Welsh, MBBS,FRCR, Principal Investigator — Royal Marsden Hospital NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stelzer KJ. Epidemiology and prognosis of brain metastases. Surg Neurol Int. 2013 May 2;4(Suppl 4):S192-202. doi: 10.4103/2152-7806.111296. Print 2013. PMID 23717790
- [Background] Lowery FJ, Yu D. Brain metastasis: Unique challenges and open opportunities. Biochim Biophys Acta Rev Cancer. 2017 Jan;1867(1):49-57. doi: 10.1016/j.bbcan.2016.12.001. Epub 2016 Dec 6. PMID 27939792
- [Background] Hoffman JM. New advances in brain tumor imaging. Curr Opin Oncol. 2001 May;13(3):148-53. doi: 10.1097/00001622-200105000-00003. PMID 11307056
- [Background] Hein PA, Eskey CJ, Dunn JF, Hug EB. Diffusion-weighted imaging in the follow-up of treated high-grade gliomas: tumor recurrence versus radiation injury. AJNR Am J Neuroradiol. 2004 Feb;25(2):201-9. PMID 14970018
- [Background] Sundgren PC, Fan X, Weybright P, Welsh RC, Carlos RC, Petrou M, McKeever PE, Chenevert TL. Differentiation of recurrent brain tumor versus radiation injury using diffusion tensor imaging in patients with new contrast-enhancing lesions. Magn Reson Imaging. 2006 Nov;24(9):1131-42. doi: 10.1016/j.mri.2006.07.008. Epub 2006 Sep 18. PMID 17071335
- [Background] Matsusue E, Fink JR, Rockhill JK, Ogawa T, Maravilla KR. Distinction between glioma progression and post-radiation change by combined physiologic MR imaging. Neuroradiology. 2010 Apr;52(4):297-306. doi: 10.1007/s00234-009-0613-9. Epub 2009 Oct 16. PMID 19834699
- [Background] Rock JP, Scarpace L, Hearshen D, Gutierrez J, Fisher JL, Rosenblum M, Mikkelsen T. Associations among magnetic resonance spectroscopy, apparent diffusion coefficients, and image-guided histopathology with special attention to radiation necrosis. Neurosurgery. 2004 May;54(5):1111-7; discussion 1117-9. doi: 10.1227/01.neu.0000119328.56431.a7. PMID 15113465
- [Background] Zach L, Guez D, Last D, Daniels D, Grober Y, Nissim O, Hoffmann C, Nass D, Talianski A, Spiegelmann R, Tsarfaty G, Salomon S, Hadani M, Kanner A, Blumenthal DT, Bukstein F, Yalon M, Zauberman J, Roth J, Shoshan Y, Fridman E, Wygoda M, Limon D, Tzuk T, Cohen ZR, Mardor Y. Delayed contrast extravasation MRI: a new paradigm in neuro-oncology. Neuro Oncol. 2015 Mar;17(3):457-65. doi: 10.1093/neuonc/nou230. Epub 2014 Nov 30. PMID 25452395
- [Background] Chen K, Chen X. Positron emission tomography imaging of cancer biology: current status and future prospects. Semin Oncol. 2011 Feb;38(1):70-86. doi: 10.1053/j.seminoncol.2010.11.005. PMID 21362517
- [Background] Nanni C, Rubello D, Fanti S. Could choline PET play a role in malignancies other than prostate cancer? Eur J Nucl Med Mol Imaging. 2008 Jan;35(1):216-8. doi: 10.1007/s00259-007-0591-2. Epub 2007 Sep 26. No abstract available. PMID 17899074
- [Background] Zeisel SH, Blusztajn JK. Choline and human nutrition. Annu Rev Nutr. 1994;14:269-96. doi: 10.1146/annurev.nu.14.070194.001413. PMID 7946521
- [Background] Fagone P, Jackowski S. Phosphatidylcholine and the CDP-choline cycle. Biochim Biophys Acta. 2013 Mar;1831(3):523-32. doi: 10.1016/j.bbalip.2012.09.009. Epub 2012 Sep 23. PMID 23010477
- [Background] Treglia G, Sadeghi R, Del Sole A, Giovanella L. Diagnostic performance of PET/CT with tracers other than F-18-FDG in oncology: an evidence-based review. Clin Transl Oncol. 2014 Sep;16(9):770-5. doi: 10.1007/s12094-014-1168-8. Epub 2014 Mar 20. PMID 24647843
- [Background] Treglia G, Giovannini E, Di Franco D, Calcagni ML, Rufini V, Picchio M, Giordano A. The role of positron emission tomography using carbon-11 and fluorine-18 choline in tumors other than prostate cancer: a systematic review. Ann Nucl Med. 2012 Jul;26(6):451-61. doi: 10.1007/s12149-012-0602-7. Epub 2012 May 8. PMID 22566040
- [Background] Kato T, Shinoda J, Nakayama N, Miwa K, Okumura A, Yano H, Yoshimura S, Maruyama T, Muragaki Y, Iwama T. Metabolic assessment of gliomas using 11C-methionine, [18F] fluorodeoxyglucose, and 11C-choline positron-emission tomography. AJNR Am J Neuroradiol. 2008 Jun;29(6):1176-82. doi: 10.3174/ajnr.A1008. Epub 2008 Apr 3. PMID 18388218
- [Background] Ohtani T, Kurihara H, Ishiuchi S, Saito N, Oriuchi N, Inoue T, Sasaki T. Brain tumour imaging with carbon-11 choline: comparison with FDG PET and gadolinium-enhanced MR imaging. Eur J Nucl Med. 2001 Nov;28(11):1664-70. doi: 10.1007/s002590100620. PMID 11702108
- [Background] Tian M, Zhang H, Oriuchi N, Higuchi T, Endo K. Comparison of 11C-choline PET and FDG PET for the differential diagnosis of malignant tumors. Eur J Nucl Med Mol Imaging. 2004 Aug;31(8):1064-72. doi: 10.1007/s00259-004-1496-y. Epub 2004 Mar 11. PMID 15014903
- [Background] Gao L, Xu W, Li T, Zheng J, Chen G. Accuracy of 11C-choline positron emission tomography in differentiating glioma recurrence from radiation necrosis: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Jul;97(29):e11556. doi: 10.1097/MD.0000000000011556. PMID 30024551
- [Background] Li Y, Jin G, Su D. Comparison of Gadolinium-enhanced MRI and 18FDG PET/PET-CT for the diagnosis of brain metastases in lung cancer patients: A meta-analysis of 5 prospective studies. Oncotarget. 2017 May 30;8(22):35743-35749. doi: 10.18632/oncotarget.16182. PMID 28415747
- [Background] Li H, Deng L, Bai HX, Sun J, Cao Y, Tao Y, States LJ, Farwell MD, Zhang P, Xiao B, Yang L. Diagnostic Accuracy of Amino Acid and FDG-PET in Differentiating Brain Metastasis Recurrence from Radionecrosis after Radiotherapy: A Systematic Review and Meta-Analysis. AJNR Am J Neuroradiol. 2018 Feb;39(2):280-288. doi: 10.3174/ajnr.A5472. Epub 2017 Dec 14. PMID 29242363
- [Background] Wagner S, Lanfermann H, Eichner G, Gufler H. Radiation injury versus malignancy after stereotactic radiosurgery for brain metastases: impact of time-dependent changes in lesion morphology on MRI. Neuro Oncol. 2017 Apr 1;19(4):586-594. doi: 10.1093/neuonc/now193. PMID 27634933
- [Background] Treglia G, Muoio B, Trevisi G, Mattoli MV, Albano D, Bertagna F, Giovanella L. Diagnostic Performance and Prognostic Value of PET/CT with Different Tracers for Brain Tumors: A Systematic Review of Published Meta-Analyses. Int J Mol Sci. 2019 Sep 20;20(19):4669. doi: 10.3390/ijms20194669. PMID 31547109
- [Background] National Instituite for Health Care and Excellence. Brain tumours (primary) and brain metastases in adults. NICE Guidel NG99. 2018;(July):1-56.
- [Background] NHS England. D05/S/a NHS STANDARD CONTRACT FOR STEREOTACTIC RADIOSURGERY AND STEREOTACTIC RADIOTHERAPY (INTRACRANIAL) (ALL AGES) SCHEDULE 2- THE SERVICES - A. SERVICE SPECIFICATIONS. 2013;800(October):1-26.